CLINICAL TRIAL: NCT05537792
Title: User-Independent Intent Recognition on a Powered Transfemoral Prosthesis
Brief Title: Intent Recognition for Prosthesis Control
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia Institute of Technology (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: H21117; DP2HD111709 (NIH)
Record Dates: First submitted 2022-09-08; First posted 2022-09-13 (Actual); Results first posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-08

CONDITIONS: Amputation
Keywords: Protheses; Amputation

STUDY DESIGN:
Intervention Model Description: The model used is a repeated measures single arm study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Smart Robotic Knee/Ankle Prothesis (Experimental): This study will be conducted on a sample population of individuals with transfemoral amputation (single arm). Each participant will test with each condition of the study (repeated measures).
  Interventions: Device: Robotic Knee/Ankle Prosthesis

INTERVENTIONS:
Device: Robotic Knee/Ankle Prosthesis — The intervention is an experimental robotic knee/ankle prosthesis that has been previously developed by the team. It is used to improve walking gait performance.

SUMMARY:
This work will focus on new algorithms for powered prostheses and testing these in human subject tests. Individuals with above knee amputation will walk with a robotic prosthesis and ambulate over terrain that simulates community ambulation. The investigators will compare the performance of the advanced algorithm with the robotic system that does not use an advanced algorithm.

DETAILED DESCRIPTION:
The focus of this work is a proposed novel AI system to self-adapt an intent recognition system in powered prostheses to aid deployment of intent recognition systems that personalize to individual patient gait. The investigators hypothesize that the prosthesis using our self-adaptive intent recognition system will improve walking speed. Independent community ambulation is known to be more challenging for individuals with TFA, and so the investigators will measure self-selected walking speed (SSWS) which is a correlate with overall health and is a predictor of functional dependence, mobility disability and falls; furthermore, slow SSWS are correlated to lower quality of life (QOL), decreased participation and symptoms of depression. Self-adapting intent recognition has great potential to restore gait in community settings and improve embodiment, which has been associated with improved QOL and increased device usage in patients who use advanced upper limb prostheses. In this experiment, patients with TFA will be fit with our robotic knee/ankle prosthesis and proceed to walk over a treadmill and overground at varying speeds, while the investigators capture 3D biomechanics in both the self-adaptive and static user-independent system (control condition). The investigators expect the self-adaptive system to learn the best prediction of the patient's unique gait, leading to advantages in functional and patient reported outcomes over the control and baseline conditions.

ELIGIBILITY:
Inclusion Criteria:

* A unilateral amputation of the lower limb
* Aged between 18 to 75 years, inclusive
* K3 or K4 level ambulators who can perform all locomotor tasks of interest (based on assessment of the physiatrist and/or prosthetist)
* If a prosthesis is used, the participant must use a prosthetic knee and foot in their clinically prescribed prosthesis.

Exclusion Criteria:

* Individuals with history of neurological injury, gait pathology, or cardiovascular condition that would limit ability to ambulate for multiple hours
* Individuals who are currently pregnant (based on patient self-report) due to slight risk of falling during experiments

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Young, Ph.D., Principal Investigator — Georgia Institute of Technology
Locations (1):
- Exoskeleton and Prosthetic Intelligent Controls Lab, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Smart Robotic Knee/Ankle Prothesis
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Smart Robotic Knee/Ankle Prothesis
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.4 (12.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
Height [Mean (Standard Deviation); unit: Meters] | 1.69 (0.10)
Weight [Mean (Standard Deviation); unit: Kilograms] | 71.83 (14.66)
Amputated Side [Count of Participants; unit: Participants]
  Amputated Side Right | 6
  Amputated Side Left | 4

OUTCOME MEASURES:

1. Primary Outcome: Overground Self-selected Walking Speed
Description: This measures the individuals preferred overground walking speed which indicates their physical capability with a device.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Meters per second
Arm/Group | Smart Robotic Knee/Ankle Prothesis
Number analyzed (Participants) | 10
Meters per second | 0.695 (0.136)

2. Secondary Outcome: Overground Walking Speed Mean Absolute Error (MAE)
Description: This outcome is the error with which the machine learning model embedded into our advanced prosthesis controller's microprocessor predicts the user's walking speed overground. Specifically, mean absolute error (MAE) is computed between the predicted walking speed and the ground truth walking speed, or the speed that the user is actually walking at. Ground truth measurements are measured by a motion-capture system and taken to be center of mass speed. Walking speed predictions are made every 50 ms and compared to the nearest center-of-mass speed. For this measure, lower walking speed MAEs are indicative of greater accuracy in defining the user's true walking speed and thus lower numbers are indicative of an improved outcome.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Mean Absolute Error for Meter per second
Arm/Group | Smart Robotic Knee/Ankle Prothesis
Number analyzed (Participants) | 10
Mean Absolute Error for Meter per second | 0.142 (0.035)

3. Secondary Outcome: Treadmill Walking Speed Mean Absolute Error (MAE)
Description: This outcome is the error with which the machine learning model embedded into our advanced prosthesis controller's microprocessor predicts the user's walking speed on the treadmill. Specifically, mean absolute error (MAE) is computed between the predicted walking speed and the ground truth walking speed, or the speed that the user is actually walking at. Ground truth measurements are measured by the true treadmill speed (for treadmill trials). Walking speed predictions are made every 50 ms and compared to the nearest center-of-mass speed. For this measure, lower walking speed MAEs are indicative of greater accuracy in defining the user's true walking speed and thus lower numbers are indicative of an improved outcome.
Time Frame: 1 day
Measure: Mean (Standard Deviation); unit: Mean Absolute Error for Meter per second
Groups:
- Baseline Estimator: This study will be conducted on a sample population of individuals with transfemoral amputation. In this baseline estimator arm, each participant will test the prosthesis with a baseline control system in which the system does not adapt to the participant's own walking speed.
  Robotic Knee/Ankle Prosthesis: The intervention is an experimental robotic knee/ankle prosthesis that has been previously developed by the team. It is used to improve walking gait performance.
- Profile 1 Inertial Measurement Unit Adapted Forward Estimator: This study will be conducted on a sample population of individuals with transfemoral amputation. In the Profile 1 inertial measurement unit adapted forward estimator arm, each participant will test the prosthesis with an adapted control system using a foot inertial measurement unit with discrete treadmill speed profiles following a staircase profile. In this treadmill speed profile participants walk at discrete speeds of 0.3, 0.5, 0.7, 0.9, 0.8, 0.6, 0.4 m/s. Each speed was maintained for 20 seconds before transitioning to the next speed at an acceleration of 0.1 meters per second squared.
  Robotic Knee/Ankle Prosthesis: The intervention is an experimental robotic knee/ankle prosthesis that has been previously developed by the team. It is used to improve walking gait performance.
- Profile 1 Ground Truth Adapted Forward Estimator: This study will be conducted on a sample population of individuals with transfemoral amputation. In the Profile 1 Ground Truth arm, each participant will test the prosthesis with an adapted control system using ground truth treadmill speeds (directly read from the treadmill controller) with treadmill speed profiles following a staircase profile. In this treadmill speed profile participants walk at discrete speeds of 0.3, 0.5, 0.7, 0.9, 0.8, 0.6, 0.4 m/s. Each speed was maintained for 20 seconds before transitioning to the next speed at an acceleration of 0.1 meters per second squared.
  Robotic Knee/Ankle Prosthesis: The intervention is an experimental robotic knee/ankle prosthesis that has been previously developed by the team. It is used to improve walking gait performance.
- Profile 2 Inertial Measurement Unit Adapted Forward Estimator: This study will be conducted on a sample population of individuals with transfemoral amputation. In the Profile 2 inertial measurement unit adapted forward estimator arm, each participant will test the prosthesis with an adapted control system using a foot inertial measurement unit with treadmill speed profiles following a triangular profile such that the treadmill speed started at 0.3 m/s, accelerated to 0.9 m/s, and then decelerated back to 0.3 m/s at a rate of 0.1 meters per second squared.
  Robotic Knee/Ankle Prosthesis: The intervention is an experimental robotic knee/ankle prosthesis that has been previously developed by the team. It is used to improve walking gait performance.
  Robotic Knee/Ankle Prosthesis: The intervention is an experimental robotic knee/ankle prosthesis that has been previously developed by the team. It is used to improve walking gait performance.
- Profile 2 Ground Truth Adapted Forward Estimator: This study will be conducted on a sample population of individuals with transfemoral amputation. In the Profile 1 Ground Truth arm,each participant will test the prosthesis with an adapted control system using ground truth treadmill speeds (directly read from the treadmill controller) with treadmill speed profiles following a triangular profile such that the treadmill speed started at 0.3 m/s, accelerated to 0.9 m/s, and then decelerated back to 0.3 m/s at a rate of 0.1 meters per second squared.
  Robotic Knee/Ankle Prosthesis: The intervention is an experimental robotic knee/ankle prosthesis that has been previously developed by the team. It is used to improve walking gait performance.
Arm/Group | Baseline Estimator | Profile 1 Inertial Measurement Unit Adapted Forward Estimator | Profile 1 Ground Truth Adapted Forward Estimator | Profile 2 Inertial Measurement Unit Adapted Forward Estimator | Profile 2 Ground Truth Adapted Forward Estimator
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10
Mean Absolute Error for Meter per second | 0.158 (0.037) | 0.155 (0.038) | 0.139 (0.039) | 0.163 (0.045) | 0.138 (0.028)
Statistical Analysis 1: Comparison: Baseline Estimator vs Profile 1 Inertial Measurement Unit Adapted Forward Estimator; Test type: Other — Paired t-tests were used to compare the offline forward estimation error of each adapted forward estimator with the baseline during overground walking; p = 0.579, t-test, 1 sided
Statistical Analysis 2: Comparison: Baseline Estimator vs Profile 1 Ground Truth Adapted Forward Estimator; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.0008, t-test, 1 sided
Statistical Analysis 3: Comparison: Baseline Estimator vs Profile 2 Inertial Measurement Unit Adapted Forward Estimator; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.5513, t-test, 1 sided
Statistical Analysis 4: Comparison: Baseline Estimator vs Profile 2 Ground Truth Adapted Forward Estimator; Test type: Other — [test comment as in outcome 3, analysis 1]; p = 0.00034, t-test, 1 sided

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Smart Robotic Knee/Ankle Prothesis
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

LIMITATIONS AND CAVEATS:
A limitation of this study involved the lack of real-time adaptation and evaluation of forward estimators during overground walking. Future studies should evaluate forward estimators in real-time for longer bouts of walking.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-08-06): https://cdn.clinicaltrials.gov/large-docs/92/NCT05537792/Prot_SAP_001.pdf
  • Informed Consent Form (2024-03-15): https://cdn.clinicaltrials.gov/large-docs/92/NCT05537792/ICF_000.pdf